CLINICAL TRIAL: NCT02910739
Title: A Two-Part, Open-Label Study to Investigate the Single-Dose Pharmacokinetics of MK-8931 When Administered to Subjects With Mild and Moderate Hepatic Insufficiency
Brief Title: An Open-Label Study Investigating MK-8931 in Participants With Mild and Moderate Hepatic Insufficiency (MK-8931-016)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P08593; Celerion Project Number (Other: CA13011); Merck Protocol Number (Other: MK-8931-016)
Record Dates: First submitted 2016-09-20; First posted 2016-09-22 (Estimated); Results first posted 2018-10-01 (Actual); Last update posted 2018-10-01 (Actual); Status verified 2018-02

CONDITIONS: Amnestic Mild Cognitive Impairment; Alzheimer's Disease; Prodromal Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — verubecestat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Part I: MK-8931 40 mg in Moderate HI Participants (Experimental): Single oral dose of MK-8931 40 mg tablet in participants with moderate HI in fasted state (Part I)
  Interventions: Drug: MK-8931
- Part I: MK-8931 40 mg in Healthy Participants (Active Comparator): Single oral dose of MK-8931 40 mg tablet in healthy matched participants in fasted state (Part I)
  Interventions: Drug: MK-8931
- Part II: MK-8931 40 mg in Mild HI Participants (Experimental): Single oral dose of MK-8931 40 mg tablet in participants with mild HI in fasted state (Part II)
  Interventions: Drug: MK-8931
- Part II: MK-8931 40 mg in Healthy Participants (Active Comparator): Single oral dose of MK-8931 40 mg tablet in healthy matched participants in fasted state (Part II)
  Interventions: Drug: MK-8931

INTERVENTIONS:
Drug: MK-8931 — MK-8931 40 mg
  Other Names: Verubecestat

SUMMARY:
This study consists of Part I and an optional Part II. The purpose of Part I is to compare the plasma pharmacokinetics of verubecestat (MK-8931) following administration of a single oral dose of 40 mg MK-8931 to participants with moderate hepatic insufficiency (HI) to that of healthy matched controls. An interim safety and pharmacokinetic analysis on the basis of Part I will be performed in order to support the decision to continue with the optional Part II. If a decision to continue with Part II is made, participants with mild HI will be enrolled to receive a single oral dose of 40mg MK-8931. If any healthy participants from Part I do not meet the matching criteria for Part II additional healthy participants will be enrolled.

ELIGIBILITY:
Inclusion Criteria: Participants with HI

1. Adult male or female participants, 45-85 years of age, inclusive, at screening.
2. Body Mass Index (BMI) ≥ 19 and ≤ 40 kg/m^2, at screening.
3. Continuous non-smokers or light smokers (< 10 cigarettes/day or the equivalent).
4. Baseline health is judged to be stable based on medical history (except for the hepatic insufficiency condition).
5. Participant has a diagnosis of chronic (> 6 months), stable (no acute episodes of illness within the previous 2 months due to deterioration in hepatic function) HI with features of cirrhosis due to any etiology.
6. Part 1 only: Participant's score on the Child-Pugh scale must range from 7 to 9 (moderate HI) at screening.
7. Part 2 only: Participant's score on the Child-Pugh scale must range from 5 to 6 (mild HI) at screening.
8. Participants must be completely informed of the unknown risks of pregnancy and agree not to become pregnant or father a child during the time they are participating in this study.
9. For a female of childbearing potential: either be sexually inactive (abstinent) for 14 days prior to dosing and throughout the study or be using an acceptable birth control method.
10. Females of non-childbearing potential must have undergone one of the following sterilization procedures at least 6 months prior to the first dose:

    * hysteroscopic sterilization;
    * bilateral tubal ligation or bilateral salpingectomy;
    * hysterectomy;
    * bilateral oophorectomy; or be postmenopausal with amenorrhea for at least 1 year prior to dosing and have follicle-stimulating hormone (FSH) serum levels consistent with postmenopausal status as per Investigator or designee's judgment.
11. Non-vasectomized male participants must agree to use a condom with spermicide or abstain from sexual intercourse from dosing until 90 days after dosing.
12. Male participants must agree not to donate sperm from dosing until 90 days after dosing.
13. Understands the study procedures in informed consent forms (ICFs), be willing and able to comply with the protocol, and provides written informed consent for the trial, including for Future Biomedical Research. Future Biomedical Research participation is voluntary and is not required in order to participate in the trial.

Inclusion Criteria: Healthy Control Participants

1. Healthy adult male or female participants, 45-85 years of age, inclusive, at screening.
2. BMI ≥ 19 and ≤ 40 kg/m^2 at screening.
3. Continuous non-smokers or light smokers (< 10 cigarettes/day or the equivalent).
4. Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs, or electrocardiograms (ECGs), as deemed by the Investigator.
5. Participants must be completely informed of the unknown risks of pregnancy and agree not to become pregnant or father a child during the time they are participating in this study.
6. For a female of childbearing potential: either be sexually inactive (abstinent) for 14 days prior to dosing and throughout the study or be using an acceptable birth control method.
7. Females of non-childbearing potential must have undergone one of the following sterilization procedures at least 6 months prior to the first dose:

   * hysteroscopic sterilization;
   * bilateral tubal ligation or bilateral salpingectomy;
   * hysterectomy;
   * bilateral oophorectomy; or be postmenopausal with amenorrhea for at least 1 year prior to dosing and have FSH serum levels consistent with postmenopausal status as per Investigator or designee's judgment.
8. Non-vasectomized male participants must agree to use a condom with spermicide or abstain from sexual intercourse from dosing until 90 days after dosing.
9. Male participants must agree not to donate sperm from dosing until 90 days after dosing.
10. Understands the study procedures in ICFs, be willing and able to comply with the protocol, and provides written informed consent for the trial, including for Future Biomedical Research. Future Biomedical Research participation is voluntary and is not required in order to participate in the trial.

Exclusion Criteria: Participants with HI

1. Participant is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
2. History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the Investigator.
3. History of any illness that, in the opinion of the Investigator, might confound the results of the study or poses an additional risk to the participant by their participation in the study.
4. History or presence of alcoholism or drug abuse within the past 2 years prior to dosing.
5. History or presence of hypersensitivity or idiosyncratic reaction to the study drug or related compounds.
6. Female participants who are pregnant or lactating.
7. Positive results for the urine drug and/or alcohol screen at screening or check-in, unless the positive drug screen is due to prescription drug use and is approved by the Investigator and the Sponsor Medical Monitor.
8. Positive results at screening for human immunodeficiency virus (HIV) or hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV; i.e., HCV antibody positive, HCV ribonucleic acid (RNA) positive) with decompensated liver disease.
9. Seated blood pressure is less than 90/40 mmHg or greater than 180/105 mmHg at screening.
10. Seated heart rate is lower than 40 bpm or higher than 99 bpm at screening.
11. Fridericia's correction of the QT interval (QTcF) is > 480 msec or has ECG findings deemed abnormal with clinical significance by the Investigator or designee at screening.
12. Abnormal hemoglobin level deemed clinically significant by the Investigator at screening.
13. Unable to refrain from or anticipates the use of any medication or substance (including prescription or over-the-counter, vitamin supplements, natural or herbal supplements).
14. Has been on a diet incompatible with the Clinical Research Unit (CRU) -provided standard meals/snacks, in the opinion of the Investigator, within the 28 days prior to dosing of study drug, and throughout the study.
15. Donation of blood or had significant blood loss within 56 days prior to dosing of study drug.
16. Plasma donation within 28 days prior to dosing of study drug.
17. Is or has an immediate family member (e.g., spouse, parent/legal guardian, sibling or child) who is investigational site or Sponsor staff directly involved with this study.
18. Participation in another clinical trial within 28 days prior to dosing.
19. Participant who dosed in one part (e.g., Part 1) will not be enrolled in the other part (e.g., Part 2).

Exclusion Criteria: Healthy Control Participants

1. Participant is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
2. History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the Investigator.
3. History of any illness that, in the opinion of the Investigator, might confound the results of the study or poses an additional risk to the participant by their participation in the study.
4. History or presence of alcoholism or drug abuse within the past 2 years prior to dosing.
5. History or presence of hypersensitivity or idiosyncratic reaction to the study drug or related compounds.
6. Female participants who are pregnant or lactating.
7. Positive results for the urine drug and/or urine or breath alcohol screen at screening or check-in.
8. Positive results at screening for HIV or HBsAg or HCV with decompensated liver disease.
9. Seated blood pressure is less than 90/40 mmHg or greater than 140/90 mmHg at screening.
10. Seated heart rate is lower than 40 bpm or higher than 99 bpm at screening.
11. QTcF is > 480 msec or has ECG findings deemed abnormal with clinical significance by the Investigator or designee at screening.
12. Abnormal hemoglobin level deemed clinically significant by the Investigator at screening.
13. Unable to refrain from or anticipates the use of any medication or substance (including prescription or over-the-counter, vitamin supplements, natural or herbal supplements).
14. Has been on a diet incompatible with the CRU-provided standard meals/snacks, in the opinion of the Investigator, within the 28 days prior to dosing of study drug, and throughout the study.
15. Donation of blood or had significant blood loss within 56 days prior to dosing of study drug.
16. Plasma donation within 28 days prior to dosing of study drug.
17. Is or has an immediate family member (e.g., spouse, parent/legal guardian, sibling or child) who is investigational site or Sponsor staff directly involved with this study.
18. Participation in another clinical trial within 28 days prior to dosing.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-10-11 (Actual); Primary Completion 2017-04-03 (Actual); Study Completion 2017-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Per protocol, this study was divided into Part I and an optional Part II, with Part II initiating only after interim analysis (IA) of Part I. Following Part I IA, the pharmacokinetic (PK) criterion necessary to initiate enrollment for Part II was not met. As a result, the study was completed normally without enrollment into the optional Part II.
Groups:
- Part I: MK-8931 40 mg in Moderate HI Participants: Single oral dose of MK-8931 (40 mg tablet) in participants with moderate Hepatic Insufficiency (HI) in fasted state (Part I)
- Part I: MK-8931 40 mg in Healthy Participants: Single oral dose of MK-8931 (40 mg tablet) in healthy matched participants in fasted state (Part I)
- Part II: MK-8931 40 mg in Mild HI Participants: Single oral dose of MK-8931 (40 mg tablet) in participants with mild HI in fasted state (Part II)
- Part II: MK-8931 40 mg in Healthy Participants: Single oral dose of MK-8931 (40 mg tablet) in healthy matched participants in fasted state (Part II)
Period: Overall Study
Arm/Group | Part I: MK-8931 40 mg in Moderate HI Participants | Part I: MK-8931 40 mg in Healthy Participants | Part II: MK-8931 40 mg in Mild HI Participants | Part II: MK-8931 40 mg in Healthy Participants
Started | 8 | 8 | 0 (Participants were not enrolled in Part II as the PK criterion from the Part I IA was not met.) | 0 (Participants were not enrolled in Part II as the PK criterion from the Part I IA was not met.)
Completed | 7 | 8 | 0 (Participants were not enrolled in Part II as the PK criterion from the Part I IA was not met.) | 0 (Participants were not enrolled in Part II as the PK criterion from the Part I IA was not met.)
Not Completed | 1 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part I: MK-8931 40 mg in Moderate HI Participants: Single oral dose of MK-8931 (40 mg tablet) in participants with moderate HI in fasted state (Part I)
- Total: Total of all reporting groups
Arm/Group | Part I: MK-8931 40 mg in Moderate HI Participants | Part I: MK-8931 40 mg in Healthy Participants | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (6.1) | 61.4 (4.8) | 61.2 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 7 | 7 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 7 | 7 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Full Range); unit: kg/m^2] | 29.688 [20.40 to 36.10] | 30.313 [27.50 to 32.60] | 30.000 [20.40 to 36.10]

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration Versus Time Curve of MK-8931 From 0 to Infinity (AUC0-∞)
Description: Blood samples were collected at each pre-specified time point and plasma was isolated for analysis. Plasma MK-8931 concentration was then quantified at each time point to determine AUC0-∞, defined as the area under the MK-8931 concentration versus time curve from 0 (predose) extrapolated to infinity after a single oral dose of MK-8931 40 mg. Individual AUC0-∞ values were natural log (ln) transformed and evaluated with an analysis of covariance (ANCOVA) model containing a categorical factor for participant group (Moderate HI, Healthy Matched Control) and continuous covariates for age and BMI. This ANCOVA model was used to compute a geometric least-squares mean and 95% confidence interval for AUC0-∞ in each arm.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, and 120 hours after MK-8931 40 mg dose
Population: All participants who received the single dose of MK-8931 40 mg, complied with trial protocol, and had blood samples available for the evaluation of AUC0-∞. One participant with moderate HI discontinued study prior to collection of samples at 72, 96, and 120 hours post-dose and was excluded from analysis.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: micromolar(µM)*hour(hr)
Arm/Group | Part I: MK-8931 40 mg in Moderate HI Participants | Part I: MK-8931 40 mg in Healthy Participants
Number analyzed (Participants) | 7 | 8
micromolar(µM)*hour(hr) | 3.48 [2.85 to 4.25] | 3.34 [2.77 to 4.03]
Statistical Analysis 1: Comparison: Part I: MK-8931 40 mg in Moderate HI Participants vs Part I: MK-8931 40 mg in Healthy Participants; Per study protocol, the purpose of this analysis is only to estimate the effect of moderate HI on AUC0-∞; no hypothesis testing was planned for this outcome measure; Test type: Other — The pharmacokinetic condition to initiate Part 2 of the study would be met if the point estimate for the AUC0-∞ ratio of geometric means (participants with moderate HI / healthy matched control participants) exceeds 1.5; Geometric least-squares mean ratio (GMR) = 1.04, 90% CI 2-sided [0.83 to 1.30] — GMR = geometric least squares mean (GLSM) for moderate HI participants / GLSM for healthy participants

2. Primary Outcome: Maximum Observed Plasma Concentration of MK-8931 (Cmax)
Description: Blood samples were collected at each pre-specified time point and plasma was isolated for analysis. Plasma MK-8931 concentration was then quantified at each time point to determine Cmax, defined as the maximum plasma concentration of MK-8931 observed following oral dosing. Individual Cmax values were ln-transformed and evaluated with an ANCOVA model containing a categorical factor for participant group (Moderate HI, Healthy Matched Control) and continuous covariates for age and BMI. This ANCOVA model was used to compute a geometric least-squares mean and 95% confidence interval for Cmax in each arm.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, and 48 hours after MK-8931 40 mg dose
Population: All participants who received the single dose of MK-8931 40 mg, complied with trial protocol, and had blood samples available for the evaluation of Cmax.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: nanomolar (nM)
Arm/Group | Part I: MK-8931 40 mg in Moderate HI Participants | Part I: MK-8931 40 mg in Healthy Participants
Number analyzed (Participants) | 8 | 8
nanomolar (nM) | 154 [116 to 206] | 144 [108 to 192]
Statistical Analysis 1: Comparison: Part I: MK-8931 40 mg in Moderate HI Participants vs Part I: MK-8931 40 mg in Healthy Participants; Per study protocol, the purpose of this analysis is only to estimate the effect of moderate HI on Cmax; no hypothesis testing was planned for this outcome measure; Test type: Other; GMR = 1.07, 90% CI 2-sided [0.77 to 1.50] — GMR = GLSM for moderate HI participants / GLSM for healthy participants

3. Primary Outcome: Area Under the Concentration Versus Time Curve of MK-8931 From 0 to the Time of the Last Quantifiable (Above LLOQ) Sample (AUC0-last)
Description: Blood samples were collected at each pre-specified time point and plasma was isolated for analysis. Plasma MK-8931 concentration was then quantified at each time point to determine AUC0-last, defined as the area under the MK-8931 concentration versus time curve from 0 (predose) to the time of the last sample with quantifiable MK-8931 (above the lower limit of quantification; LLOQ) after a single oral dose of MK-8931 40 mg. Individual AUC0-last values were ln-transformed and evaluated with an ANCOVA model containing a categorical factor for participant group (Moderate HI, Healthy Matched Control) and continuous covariates for age and BMI. This ANCOVA model was used to compute a geometric least-squares mean and 95% confidence interval for AUC0-last in each arm.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, and 120 hours after MK-8931 40 mg dose
Population: All participants who received the single dose of MK-8931 40 mg, complied with trial protocol, and had blood samples available for the evaluation of AUC0-last. One participant with moderate HI discontinued study prior to collection of samples at 72, 96, and 120 hours post-dose and was excluded from analysis.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: µM*hr
Arm/Group | Part I: MK-8931 40 mg in Moderate HI Participants | Part I: MK-8931 40 mg in Healthy Participants
Number analyzed (Participants) | 7 | 8
µM*hr | 3.35 [2.72 to 4.11] | 3.22 [2.66 to 3.91]
Statistical Analysis 1: Comparison: Part I: MK-8931 40 mg in Moderate HI Participants vs Part I: MK-8931 40 mg in Healthy Participants; Per study protocol, the purpose of this analysis is only to estimate the effect of moderate HI on AUC0-last; no hypothesis testing was planned for this outcome measure; Test type: Other; GMR = 1.04, 90% CI 2-sided [0.82 to 1.31] — GMR = GLSM for moderate HI participants / GLSM for healthy participants

4. Primary Outcome: Area Under the Concentration Versus Time Curve of MK-8931 From 0 to 24 Hours (AUC0-24hr)
Description: Blood samples were collected at each pre-specified time point and plasma was isolated for analysis. Plasma MK-8931 concentration was then quantified at each time point to determine AUC0-24hr, defined as the area under the MK-8931 concentration versus time curve from 0 (predose) until 24 hours after single oral dosing of MK-8931 40 mg. Individual AUC0-24hr values were ln-transformed and evaluated with an ANCOVA model containing a categorical factor for participant group (Moderate HI, Healthy Matched Control) and continuous covariates for age and BMI. This ANCOVA model was used to compute a geometric least-squares mean and 95% confidence interval for AUC0-24hr in each arm.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 hours after MK-8931 40 mg dose
Population: All participants who received the single dose of MK-8931 40 mg, complied with trial protocol, and had blood samples available for the evaluation of AUC0-24hr.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: µM*hr
Arm/Group | Part I: MK-8931 40 mg in Moderate HI Participants | Part I: MK-8931 40 mg in Healthy Participants
Number analyzed (Participants) | 8 | 8
µM*hr | 1.90 [1.56 to 2.32] | 1.88 [1.54 to 2.30]
Statistical Analysis 1: Comparison: Part I: MK-8931 40 mg in Moderate HI Participants vs Part I: MK-8931 40 mg in Healthy Participants; Per study protocol, the purpose of this analysis is only to estimate the effect of moderate HI on AUC0-24hr; no hypothesis testing was planned for this outcome measure; Test type: Other; GMR = 1.01, 90% CI 2-sided [0.80 to 1.27] — GMR = GLSM for moderate HI participants / GLSM for healthy participants

5. Primary Outcome: Plasma Concentration of MK-8931 at 24 Hours (C24hr)
Description: Blood samples were collected 24 hours following oral dosing of MK-8931 and plasma was isolated for analysis. Plasma MK-8931 concentration was then quantified to determine C24hr, defined as the plasma concentration of MK-8931 at 24 hours after single oral dosing of MK-8931 40 mg. Individual C24hr values were ln-transformed and evaluated with an ANCOVA model containing a categorical factor for participant group (Moderate HI, Healthy Matched Control) and continuous covariates for age and BMI. This ANCOVA model was used to compute a geometric least-squares mean and 95% confidence interval for C24hr in each arm.
Time Frame: 24 hours after MK-8931 40 mg dose
Population: All participants who received the single dose of MK-8931 40 mg, complied with trial protocol, and had blood samples available for the evaluation of C24hr.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: nM
Arm/Group | Part I: MK-8931 40 mg in Moderate HI Participants | Part I: MK-8931 40 mg in Healthy Participants
Number analyzed (Participants) | 8 | 8
nM | 51.1 [43.6 to 59.8] | 47.1 [40.2 to 55.2]
Statistical Analysis 1: Comparison: Part I: MK-8931 40 mg in Moderate HI Participants vs Part I: MK-8931 40 mg in Healthy Participants; Per study protocol, the purpose of this analysis is only to estimate the effect of moderate HI on C24hr; no hypothesis testing was planned for this outcome measure; Test type: Other; GMR = 1.08, 90% CI 2-sided [0.90 to 1.30] — GMR = GLSM for moderate HI participants / GLSM for healthy participants

6. Primary Outcome: Apparent Clearance of MK-8931 After Extravascular Administration (CL/F)
Description: Geometric mean apparent clearance of MK-8931 after extravascular administration (CL/F) was assessed. Blood samples were collected at each pre-specified time point and plasma was isolated for analysis. Plasma MK-8931 concentration was then quantified at each time point to determine CL/F, defined as the rate of MK-8931 elimination normalized to the bioavailability of MK-8931 in the plasma following oral MK-8931 administration.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, and 120 hours after MK-8931 40 mg dose
Population: All participants who received the single dose of MK-8931 40 mg, complied with trial protocol, and had blood samples available for the evaluation of CL/F. One participant with moderate HI discontinued study prior to collection of samples at 72, 96, and 120 hours post-dose and was excluded from analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters/hr
Arm/Group | Part I: MK-8931 40 mg in Moderate HI Participants | Part I: MK-8931 40 mg in Healthy Participants
Number analyzed (Participants) | 7 | 8
Liters/hr | 28.4 (26.3) | 29.0 (22.7)

7. Primary Outcome: Time to Maximum Observed MK-8931 Plasma Drug Concentration (Tmax)
Description: Median time to maximum observed MK-8931 plasma drug concentration (Tmax) was assessed. Blood samples were collected at each pre-specified time point and plasma was isolated for analysis. Plasma MK-8931 concentration was then quantified at each time point to determine Tmax, defined as the amount of time required following MK-8931 administration for the plasma concentration of MK-8931 to reach maximum observed concentration.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, and 48 hours after MK-8931 40 mg dose
Population: All participants who received the single dose of MK-8931 40 mg, complied with trial protocol, and had blood samples available for the evaluation of Tmax.
Measure: Median (Full Range); unit: hr
Arm/Group | Part I: MK-8931 40 mg in Moderate HI Participants | Part I: MK-8931 40 mg in Healthy Participants
Number analyzed (Participants) | 8 | 8
hr | 1.00 [0.50 to 4.00] | 2.00 [0.50 to 4.00]

8. Primary Outcome: Apparent Terminal Half-Life of MK-8931 (t1/2)
Description: Geometric mean apparent terminal half-life (t1/2) of MK-8931 was assessed. Blood samples were collected at each pre-specified time point and plasma was isolated for analysis. Plasma MK-8931 concentration was then quantified at each time point to determine t1/2, defined as the time required for the plasma MK-8931 concentration to decrease to 50% of maximum.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, and 120 hours after MK-8931 40 mg dose
Population: All participants who received the single dose of MK-8931 40 mg, complied with trial protocol, and had blood samples available for the evaluation of t1/2. One participant with moderate HI discontinued study prior to collection of samples at 72, 96, and 120 hours post-dose and was excluded from analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Part I: MK-8931 40 mg in Moderate HI Participants | Part I: MK-8931 40 mg in Healthy Participants
Number analyzed (Participants) | 7 | 8
hr | 23.0 (15.7) | 24.7 (9.3)

9. Primary Outcome: Apparent Volume of Distribution of MK-8931 During the Terminal Phase After Extravascular Administration (Vz/F)
Description: Geometric mean apparent volume of distribution of MK-8931 during the terminal phase after extravascular administration (Vz/F) was assessed. Blood samples were collected at each pre-specified time point and plasma was isolated for analysis. Plasma MK-8931 concentration was then quantified at each time point to determine Vz/F, defined as the total amount of MK-8931 administered normalized to the bioavailability of MK-8931 in the plasma during the terminal phase following oral MK-8931 administration.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, and 120 hours after MK-8931 40 mg dose
Population: All participants who received the single dose of MK-8931 40 mg, complied with trial protocol, and had blood samples available for the evaluation of Vz/F. One participant with moderate HI discontinued study prior to collection of samples at 72, 96, and 120 hours post-dose and was excluded from analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Part I: MK-8931 40 mg in Moderate HI Participants | Part I: MK-8931 40 mg in Healthy Participants
Number analyzed (Participants) | 7 | 8
Liters | 940 (27.3) | 1030 (26.1)

10. Secondary Outcome: Number of Participants Experiencing an Adverse Event
Description: The number of participants experiencing an adverse event (AE) was assessed. An AE is any unfavorable and unintended medical occurrence, symptom, or disease witnessed in a participant, regardless of whether or not a causal relationship with the study treatment can be demonstrated. Further, any worsening of a preexisting condition that is temporally associated with the use of the study treatment is also considered an AE.
Time Frame: Up to 14 days following MK-8931 40 mg administration.
Population: All participants as treated, consisting of all participants receiving the single dose of MK-8931 40 mg.
Measure: Count of Participants; unit: Participants
Arm/Group | Part I: MK-8931 40 mg in Moderate HI Participants | Part I: MK-8931 40 mg in Healthy Participants
Number analyzed (Participants) | 8 | 8
Participants | 1 | 0

11. Secondary Outcome: Number of Participants Discontinuing Study Due to an Adverse Event
Description: The number of participants discontinuing study due to an AE was assessed. An AE is any unfavorable and unintended medical occurrence, symptom, or disease witnessed in a participant, regardless of whether or not a causal relationship with the study treatment can be demonstrated. Further, any worsening of a preexisting condition that is temporally associated with the use of the study treatment is also considered an AE.
Time Frame: Up to 14 days following MK-8931 40 mg administration.
Population: All participants as treated, consisting of all participants receiving the single dose of MK-8931 40 mg.
Measure: Count of Participants; unit: Participants
Arm/Group | Part I: MK-8931 40 mg in Moderate HI Participants | Part I: MK-8931 40 mg in Healthy Participants
Number analyzed (Participants) | 8 | 8
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: Up to 14 days following MK-8931 40 mg administration.
Arm/Group | Part I: MK-8931 40 mg in Moderate HI Participants | Part I: MK-8931 40 mg in Healthy Participants
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part I: MK-8931 40 mg in Moderate HI Participants (N=8) | Part I: MK-8931 40 mg in Healthy Participants (N=8)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-05): https://cdn.clinicaltrials.gov/large-docs/39/NCT02910739/Prot_SAP_000.pdf